CLINICAL TRIAL: NCT04320095
Title: BiZact Versus Electrocautery in Tonsillectomy: A Single-Center Randomized Controlled Trial
Brief Title: Tonsillectomy Using BiZact Tonsilletomy Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB19-0088
Record Dates: First submitted 2020-03-22; First posted 2020-03-24 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Bizact device for one tonsil (Experimental): Bizact tonsillecotmy device which is an advanced bipolar device using radiofrequency and pressure to ligate the encountered vessels during tonsillectomy.
  Interventions: Device: Bizact tonsillectomy device
- Electrocautery for second tonsil (Active Comparator): Electrocautery is the standard technique used at our institution.
  Interventions: Device: Bizact tonsillectomy device
- Bizact device for both tonsils (Experimental): Consecutive cases of tonsillectomy will be done using Bizact device and compare the operative time collectively for those cases and compare it to same number of cases done using the standard procedure ( Electrocautery)
  Interventions: Device: Bizact tonsillectomy device
- Electrocautery for both tonsils (Active Comparator): As explained on the above arm description
  Interventions: Device: Bizact tonsillectomy device

INTERVENTIONS:
Device: Bizact tonsillectomy device — Bizact tonsillectomy device is an advanced bipolar instrument that uses radiofrequency energy and pressure to ligate vessels interposed between its jaws. The energy produced by the device is automatically adjusted based on tissue impedance in an attempt to minimize thermal tissue damage.

SUMMARY:
The purpose of this study is to describe how Bizact Tonsillectomy Device might affect operative time and intraoperative blood loss in pediatric patients undergoing tonsillectomy, and compare these parameters to the standard technique in tonsillectomy at our institution, which is electrocautery.

DETAILED DESCRIPTION:
It is a prospective, interventional, single-center study on the performance of Bizact tonsillectomy device on children undergoing tonsillectomy.The required parameters concerning operative time and intra operative blood loss will be obtained during the procedure.There will be no extra clinical visits for the participants.

Operative time will be assessed in 2 ways: 1). By using blade-tipped electrocautery on one tonsil and the BiZact device on the other tonsil for same patient; and 2). using electrocautery for removal of both tonsils and comparing the operative time to an equal number of cases wherein the BiZact device was used for removal of both tonsils.

With regard to intra operative bleeding, it will be quantified into one of 3 groups: 1). No blood in suction tubing, 2). blood in suction tubing but not in the suction canister, and 3). blood in the suction canister.

ELIGIBILITY:
Inclusion Criteria:

1. Children scheduled for tonsillectomy at Alberta Children Hospital
2. Tonsillectomy for either recurrent tonsillitis or sleep-disordered breathing.

Exclusion Criteria:

1. Craniofacial abnormalities
2. Bleeding disorders
3. Complex medical background

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Operative time | during the procedure
  The study will be considered success if the mean intra operative time using Bizact device is less than that using electrocautery

SECONDARY OUTCOMES:
Intraoperative blood loss | during the procedure
  The study will be considered success if the mean intraoperative blood loss using Bizact is less than Electrocautery

IPD SHARING:
Plan to Share IPD: No